CLINICAL TRIAL: NCT02497742
Title: Once Versus Twice Daily Electrolyte Monitoring in CHF; a Study Monitoring Electrolytes in Congestive Heart Failure Patients Being Actively Diuresed in Hospital
Brief Title: Once Versus Twice Daily Electrolyte Monitoring in CHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Christopher Brown, Resident Physician, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150083
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Once daily BMP (Active Comparator): Patient in this arm will receive once daily basic metabolic panel to monitor electrolytes
  Interventions: Other: Basic metabolic panel
- Twice daily BMP (Active Comparator): Patient in this arm will receive twice daily basic metabolic panel to monitor electrolytes
  Interventions: Other: Basic metabolic panel

INTERVENTIONS:
Other: Basic metabolic panel — Patients blood is collected in routine fashion for basic blood chemistries

SUMMARY:
Twice daily basic metabolic panel's or labs are common practice at Vanderbilt University Medical Center. However, it is unclear how often the second BMP each day is acted on. the investigators project aims to answer a few fundamental questions about the need for twice daily labs in patients hospitalized with acute/subacute-decompensated congestive heart failure who are being actively diuresed.

DETAILED DESCRIPTION:
Background: Over 5 million Americans are currently suffering from heart failure, resulting in over 1 million hospital admissions each year. Heart failure hospitalizations are one of the most expensive medical problems facing Americans today]. Admissions for acute decompensate heart failure exacerbations are managed medically through oral and intravenous (IV) diuretics. Side effects of diuretics are well established, the most common of which is metabolic derangements, more specifically alterations in levels of potassium . Clinical manifestations of hypokalemia and hyperkalemia are most commonly muscle cramps and clinically insignificant arrhythmia. The most concerning manifestations of hypo and hyperkalemia include symptomatic arrhythmia, myalgia, and more rarely rhabdomyolysis. Active use of diuretics requires monitoring of serum electrolytes to prevent clinically significant derangements in potassium. The frequency of monitoring required to prevent these events has not been established. Monitoring is thus provider dependent. At our single large academic medical center monitoring frequency ranges from 1-2 times daily on average. In this trial we will determine whether twice-daily electrolyte labs result in less frequent clinically hypo or hyperkalemia. We will also investigate a multitude of other outcomes including potential cost savings by reduced laboratory test ordering.

Intervention: Randomization of study population to ONCE daily scheduled BMP or TWICE daily scheduled BMP.

Risk: Risks to both arms of the study are in clinical equipoise and include: Hypokalemia, hyperkalemia, arrhythmia (secondary to hypokalemia or hyperkalemia), delayed identification of rising creatinine (acute kidney injury).

Project goals: Twice daily basic metabolic panel's or labs are common practice at Vanderbilt University Medical Center. However, it is unclear how often the second BMP each day is acted on. Our project aims to answer a few fundamental questions about the need for twice daily labs in patients hospitalized with acute/subacute-decompensated congestive heart failure who are being actively diuresed.

Descriptive:

Age Race Sex JVP on admission JVP on discharge Congestion on CXR Left ventricular ejection fraction Diabetes (Type I, or Type II [defined as HgA1C >6.5%]) Type of cardiomyopathy- ICM vs NON Ace-I or ARB Beta blocker Aldosterone antagonist HF hospitalization within past 12 months Na K (all recorded during stay) Cl BUN Cr (all recorded during stay and most recent prior to hospitalization) Total dose of loop diuretics received during admission Total dose of thiazide diuretics received Total dose of mineralocorticoid antagonist received

Outcomes:

Primary: Proportion of labs spent in ideal potassium range (defined at 3.5-5.0 mmol).

Secondary: Clinically relevant hypokalemia or hyperkalemia; defined as new muscle weakness, rhabdomyolysis, paralysis, ECG changes or conduction. Amount of potassium given, number of times per day potassium was given and average potassium value during stay. Time free from readmission, length of stay, change in weight (as surrogate for amount of diuresis), Input and output, mortality at 1mo and 3mo, cost savings during admission.

ELIGIBILITY:
Inclusion Criteria:

* Acute decompensated Heart failure (ADHF)
* actively being diuresed (home dose or greater of diuretics)
* presentation within 24 hr of enrollment
* having a history of chronic HF.

Exclusion criteria:

* First time heart failure diagnosis
* systolic blood pressure < 90mmHg
* patients requiring inotropes (other than digoxin) or milrinone
* estimated glomerular filtration rate <10.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Composite time spent in ideal potassium range | entire hospital stay, an expected average of 72 hours
  Patients average potassium during their stay will be compared to normal range defined at 3.5-5. 0 (mmol/l). , using general estimating equations allowing for comparisons between groups as well as interpersonally, in addition proportion of labs that are within normal values as stated about will also be compared between groups as well as proportion of labs in the ideal range in each group.

SECONDARY OUTCOMES:
Cost associated with hospitalization | entire hospital stay, an expected average of 72 hours
  The cost of hospitalization in each of the study arms, using ICD 9 codes billed for during the stay of hospitalization and standardized costs defined by medicare
length of stay | entire hospital stay, an expected average of 72 hours
  hospital length of stay, calculated in hours from admission to discharge
readmission rate | 1 month
  rate of readmission for congestive heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Brown, MD, Principal Investigator — Vanderbilt physician
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] 1. American Heart Association., Heart and stroke statistical update. American Heart Association: Dallas Tx. p. v.
- [Background] Ellison DH, Loffing J. Thiazide effects and adverse effects: insights from molecular genetics. Hypertension. 2009 Aug;54(2):196-202. doi: 10.1161/HYPERTENSIONAHA.109.129171. Epub 2009 Jun 29. No abstract available. PMID 19564550
- [Background] Comi G, Testa D, Cornelio F, Comola M, Canal N. Potassium depletion myopathy: a clinical and morphological study of six cases. Muscle Nerve. 1985 Jan;8(1):17-21. doi: 10.1002/mus.880080104. PMID 4058453
- [Background] Evers S, Engelien A, Karsch V, Hund M. Secondary hyperkalaemic paralysis. J Neurol Neurosurg Psychiatry. 1998 Feb;64(2):249-52. doi: 10.1136/jnnp.64.2.249. PMID 9489541
- [Background] Helfant RH. Hypokalemia and arrhythmias. Am J Med. 1986 Apr 25;80(4A):13-22. doi: 10.1016/0002-9343(86)90336-0. PMID 3706349
- [Background] Holland OB, Nixon JV, Kuhnert L. Diuretic-induced ventricular ectopic activity. Am J Med. 1981 Apr;70(4):762-8. doi: 10.1016/0002-9343(81)90530-1. PMID 7211912
- [Background] Shintani S, Shiigai T, Tsukagoshi H. Marked hypokalemic rhabdomyolysis with myoglobinuria due to diuretic treatment. Eur Neurol. 1991;31(6):396-8. doi: 10.1159/000116702. PMID 1756765
- [Background] Whelton PK. Diuretic-induced cardiac arrhythmias. Md State Med J. 1983 Dec;32(12):903-4. No abstract available. PMID 6664121
- [Background] Storrow AB, Lindsell CJ, Collins SP, Diercks DB, Filippatos GS, Hiestand BC, Hollander JE, Kirk JD, Levy PD, Miller CD, Naftilan AJ, Nowak RM, Pang PS, Peacock WF, Gheorghiade M, Cleland JG, Gheorghiade M, Abraham WT, Amsterdam EA, Cleland JG, Diercks DB, Dunlap S, Ghali J, Hobbs R, Hiestand BC, Hollander JE, Douglas Kirk J, Kremastinos D, Levy PD, Lindsell CJ, McCord J, Miller CD, Naftilan AJ, Pang PS, Frank Peacock W, Storrow AB, Thohan V. Standardized reporting criteria for studies evaluating suspected acute heart failure syndromes in the emergency department. J Am Coll Cardiol. 2012 Aug 28;60(9):822-32. doi: 10.1016/j.jacc.2012.03.072. PMID 22917006